CLINICAL TRIAL: NCT02870231
Title: A Multiple Dose Trial Investigating Safety, Tolerability, PK and PD for Multiple Doses of NNC9204-0530 in Combination With Liraglutide in Male and Female Subjects Being Overweight or With Obesity
Brief Title: Investigating Safety, Tolerability, PK and PD for Multiple Doses of NNC9204-0530 in Combination With Liraglutide in Male and Female Subjects Being Overweight or With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9030-4130; U1111-1175-7040 (Other: WHO)
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC9204-0530 / Placebo and Liraglutide 1.8 (Experimental)
  Interventions: Drug: NNC9204-0530; Drug: liraglutide; Drug: placebo
- NNC9204-0530 /Placebo and Liraglutide 3.0 (Active Comparator)
  Interventions: Drug: NNC9204-0530; Drug: liraglutide; Drug: placebo

INTERVENTIONS:
Drug: NNC9204-0530 — Once-daily subcutaneous (s.c., under the skin) administration.
Drug: liraglutide — Once-daily subcutaneous (s.c., under the skin) administration.
Drug: placebo — Once-daily subcutaneous (s.c., under the skin) administration

SUMMARY:
This trial is conducted in the United States of America. The aim of this trial is to investigate Safety, Tolerability, PK (the exposure of the trial drug in the body) and PD (the effect of the investigated drug on the body) for Multiple Doses of NNC9204-0530 in Combination with Liraglutide in Male and Female Subjects being Overweight or with Obesity

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 25.0 and 39.9 kg/m^2 (both inclusive) at screening.
* Male or female, age between 18 and 55 years (both inclusive) at the time of signing informed consent

Exclusion Criteria:

* Any clinically significant weight change (equal or above 5% self-reported change) or dieting attempts (e.g. participation in an organized weight reduction program within the last 90 days prior to screening
* Any prior obesity surgery or currently present gastrointestinal implant.
* Thyroid-stimulating hormone (TSH) values outside 0.4-6.0 mIU/L
* Glycosylated haemoglobin (HbA1c)above or equal to 6.5% or in Système International (SI) units 48 mmol/mol
* Abnormal ECG (electrocardiogram) results including 2nd or 3rd degree AV-block, prolongation of the QRS complex above 120 ms, or the QTcF interval above 430 ms (males) or above 450 ms (females), or other clinically relevant abnormal results, as judged by the investigator
* A history of additional risk factors for Torsades de pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2)
* Calcitonin above or equal to 50 ng/L
* History of pancreatitis (acute or chronic)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2017-09-03 (Actual); Study Completion 2017-09-03 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | Day 1-112

SECONDARY OUTCOMES:
Area under the NNC9204-0530 serum concentration-time curve | Day 84-112
Time to maximum serum concentration of NNC9204-0530 | Day 84-112
Change in HbA1C | Day -1, Day 85

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Novo Nordisk Investigational Site, Tempe, Arizona
  - Novo Nordisk Investigational Site, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com